CLINICAL TRIAL: NCT02693184
Title: Validation of a Revised Food Frequency Questionnaire in a Population of Elderly Men and Women With Fragility Fractures and Correlation With Bone Mineral Density and Biochemical Markers
Brief Title: Validation of a Revised Food Frequency Questionnaire
Acronym: FFQ
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0117-16-EP
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Osteoporosis; Nutrition
MeSH Terms: conditions — Osteoporosis | interventions — Vitamin D

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fragility Fracture Case: Men and women, age >65 years with a fragility fracture (defined as a fracture sustained after a fall from a standing height or less).
  Interventions: Other: Full length Block 2014 Food Frequency Questionnaire; Other: Revised Calcium, Vitamin D and Protein Screener

INTERVENTIONS:
Other: Full length Block 2014 Food Frequency Questionnaire — The food and beverage list includes 127 items, plus additional questions to adjust for fat, protein, carbohydrate, sugar, and whole grain content.
Other: Revised Calcium, Vitamin D and Protein Screener — The food list includes 29 food items and 5 supplements

SUMMARY:
The purpose of this study is to validate a revised food frequency questionnaire that is designed to capture vitamin D, calcium and protein intake in a population of elderly men and women with fragility fractures. Protein, calcium and protein intake will be correlated with biochemical measures and bone mineral density measured by DXA.

DETAILED DESCRIPTION:
The purpose of this study is to validate a revised food frequency questionnaire that is designed to capture vitamin D, calcium and protein intake in a population of elderly men and women with fragility fractures. Protein, calcium and protein intake will be correlated with biochemical measures and bone mineral density measured by DXA.

Eligibility Criteria) Forty-five eligible participants will be recruited from the endocrine referrals for osteoporosis/fracture. They will be men and women, age >65 years with a fragility fracture (defined as a fracture sustained after a fall from a standing height or less). They will be English speaking. They will need to have the mental capacity to recall events, (MMSE score ³24).11 They will need to have a telephone and the ability to answer questions over a phone. They will not have secondary causes of fragility fracture such as malabsorption (celiac disease, bariatric surgery), liver disease, organ transplant, hyperparathyroidism, multiple myeloma, current cancer diagnosis, or alcoholism. They will not have renal disease requiring dialysis (as the dietary requirement of these patients is quite different from the general elderly population). They will not be on tubefeeds of any kind (although supplemental food such as Ensure is allowed). Interventions and Evaluations) The evaluations will include a history and physical exam, and a mini mental status exam. Two telephone interviews will be conducted ~ 4 weeks apart during which the Block 2014 questionnaire will be given and the revised screener will be given. The order that the questionnaires are given will be randomized. As part of the standard of care workup for osteoporosis, a biochemical workup including 25-hydroxyvitamin D, comprehensive metabolic profile, bone specific alkaline phosphatase (a bone remodeling marker), phosphorus and transglutaminase IgA (to rule out celiac disease), and DXA scan for bone mineral density (BMD) measurement will be done. The BMD by DXA and 25-hydroxyvitamin D will be correlated to protein, calcium and vitamin D intake obtained by the Block 2014.

ELIGIBILITY:
Inclusion Criteria:

* They will be men and women, age >65 years with a fragility fracture (defined as a fracture sustained after a fall from a standing height or less). They will be English speaking. They will need to have the mental capacity to recall events, (MMSE score >24).11 They will need to have a telephone and the ability to answer questions over a phone.

Exclusion Criteria:

* They will not have secondary causes of fragility fracture such as malabsorption (celiac disease, bariatric surgery), liver disease, organ transplant, hyperparathyroidism, multiple myeloma, current cancer diagnosis, or alcoholism. They will not have renal disease requiring dialysis (as the dietary requirement of these patients is quite different from the general elderly population). They will not be on tubefeeds of any kind (although supplemental food such as Ensure is allowed).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Men and women, age >65 years with a fragility fracture (defined as a fracture sustained after a fall from a standing height or less).
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-03-25 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Agreement of the 2 FFQs on protein intake | 1 year
  Protein intake will be assessed with 2 different methods
Agreement of the 2 FFQs on calcium intake | 1 year
  Calcium intake will be assessed with 2 different methods
Agreement of the 2 FFQs on vitamin D intake | 1 year
  Vitamin D intake will be assessed with 2 different methods

CONTACTS AND LOCATIONS:
Overall Officials: Laura AG Armas, MD, MS, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
The participant will be sent a letter at the end of study detailing their calcium, protein and vitamin D intake reported on the FFQ